CLINICAL TRIAL: NCT04371250
Title: Mental Health Implications During and After the COVID-19 Pandemic Lock-down Measures in Youth (18 - 25 Years Old) in French-Speaking Belgium and Italy: Resilience and Loneliness Evaluation.
Brief Title: Study of Resilience and Loneliness in Youth (18 - 25 Years Old) During the COVID-19 Pandemic Lock-down Measures.
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Université Libre de Bruxelles (Other); King Baudouin Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2020_158
Record Dates: First submitted 2020-04-22; First posted 2020-05-01 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Resilience, Psychological; Loneliness; Youth; Surveys and Questionnaires
Keywords: Mental Health; Emerging Adulthood
MeSH Terms: conditions — Psychological Well-Being | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth: Assessed group
  Interventions: Other: Survey and Questionnaire

INTERVENTIONS:
Other: Survey and Questionnaire — Resilience and Loneliness questionnaires

SUMMARY:
The outbreak linked to SARS-CoV-2 pandemic resulted in lock-down measures in almost all European countries.

This online survey assesses these measures implications on Mental Health in emerging adults.

The questionnaires evaluate two psychometric variables (Resilience and Loneliness) and Mental Health status (mental health professional help-seeking, use of psychotropic drugs, or possible diagnosis) before and during Lock-down Measures.

At least 600 healthy participants aged form 18 to 25 years old will be attended to fill the survey during the SARS-CoV2 Pandemic Lock-down Measures.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking or Italian-speaking
* Subjects who accepted to participated to the online survey
* Inhabitants of a European country where SARS-CoV2 Pandemic Lock-down Measures are underway
* Survey filling date up to one week after the end of Lock-down Measures in the Country of residence

Exclusion Criteria:

* Incomplete surveys

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy youth living in a European Country where SARS-CoV2 Pandemic Lock-down Measures are underway.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Self-rated measure of Resilience | Up to 1 week after the end of the lock-down measures
  Measured with the Resilience Scale for Adults (RSA).
Self-rated measure of Loneliness | Up to 1 week after the end of the lock-down measures
  Measured with the UCLA (University of California, Los Angeles) Loneliness Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boffo, M., Mannarini, S., & Munari, C. (2012). Exploratory Structure Equation Modeling of the UCLA Loneliness Scale: A contribution to the Italian adaptation. TPM: Testing, Psychometrics, Methodology in Applied Psychology, 19(4).
- [Background] Bonfiglio NS, Renati R, Hjemdal O, Friborg O. The resilience scale for adults in italy: A validation study comparing clinical substance abusers with a nonclinical sample. Psychol Addict Behav. 2016 Jun;30(4):509-15. doi: 10.1037/adb0000176. Epub 2016 Mar 31. PMID 27031088
- [Background] Friborg, O., Martinussen, M., & Rosenvinge, J. H. (2006). Likert-based vs. semantic differential-based scorings of positive psychological constructs: A psychometric comparison of two versions of a scale measuring resilience. Personality and Individual Differences, 40(5), 873-884. https://doi.org/10.1016/j.paid.2005.08.015
- [Background] Grace, G. D. E., Joshi, P., Pelletier, R., & Laval, U. (1993). L'Echelle de solitude de l'Universite Laval ( ESUL ): validation canadienne-francaise du UCLA Loneliness Scale. (1959), 12-27.
- [Background] Hjemdal, O., Friborg, O., Braun, S., Kempenaers, C., Linkowski, P., & Fossion, P. (2011). The resilience scale for adults: Construct validity and measurement in a Belgian sample. International Journal of Testing, 11(1), 53-70. https://doi.org/10.1080/15305058.2010.508570
- [Background] Kessler RC, Amminger GP, Aguilar-Gaxiola S, Alonso J, Lee S, Ustun TB. Age of onset of mental disorders: a review of recent literature. Curr Opin Psychiatry. 2007 Jul;20(4):359-64. doi: 10.1097/YCO.0b013e32816ebc8c. PMID 17551351
- [Background] Marcoen A, Goossens L, Caes P. Lonelines in pre-through late adolescence: Exploring the contributions of a multidimensional approach. J Youth Adolesc. 1987 Dec;16(6):561-77. doi: 10.1007/BF02138821. PMID 24277491